CLINICAL TRIAL: NCT05960630
Title: MIRRORS-RCT (Pilot): Randomised Controlled Trial (RCT) of Robotic Interval Cytoreductive Surgery for Advanced Ovarian, Fallopian Tube and Peritoneal Cancer (EOC) Following MIRRORS-protocol vs Standard Open Interval Cytoreductive Surgery
Brief Title: MIRRORS-RCT Pilot: Role of Robotic Interval Cytoreductive Surgery for Advanced Ovarian Cancer
Acronym: MIRRORS-RCTP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Miss Christina Uwins, Sub-Speciality Fellow in Gynaecological Oncology and Associate PI, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23SURN279899
Record Dates: First submitted 2023-06-17; First posted 2023-07-27 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Ovarian Cancer; Ovarian Neoplasm; Ovarian Neoplasm Epithelial; Fallopian Tube Cancer; Fallopian Tube Neoplasms; Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIRRORS Protocol (Experimental): Diagnostic Laparoscopy proceed to either robotic or open Interval cytoreductive surgery with conversion to open at any point should this be required to remove all visible disease.
  Interventions: Procedure: MIRRORS Protocol
- Standard Care (Active Comparator): Standard Care - Open Interval Cytoreductive Surgery Surgery will proceed directly with standard open interval cytoreductive surgery through an extended midline incision
  Interventions: Procedure: Standard Open Cytoreductive Surgery

INTERVENTIONS:
Procedure: MIRRORS Protocol — Diagnostic laparoscopic assessment proceeding to either robotic (if considered appropriate following laparoscopic assessment) or open Interval cytoreductive surgery with conversion to open at any point should this be required to remove all visible disease.
  Arms: MIRRORS Protocol
Procedure: Standard Open Cytoreductive Surgery — Extended midline incision. Open surgical approach to interval cytoreductive surgery with the aim of removing all visible disease.
  Arms: Standard Care

SUMMARY:
The survival of ovarian cancer patients is dependent on the stage at diagnosis; more than 70% of patients present with advanced stage disease (stage III/IV). In England, one-year survival is 98.7% at stage I and 51.4% at stage IV and five-year survival is 93.3% and 13.4% respectively. Standard treatment for advanced ovarian cancer involves surgery to remove all visible tumour and chemotherapy. Removal of all visible disease, so no tumour deposits are visible to the naked eye at the end of first-line surgery, is one of the strongest predictors of overall survival.

A majority of the women presenting with advanced disease are older and frail. Extensive open surgery discriminates against such women as they may not be well enough for the surgery offered. A recent national audit in England found that 60.1% of women over the age of 79yrs diagnosed with ovarian cancer received no cancer treatment at all. The ability to provide the same surgery via a minimally invasive route such as robotic surgery potentially widens access to cancer treatment.

The MIRRORS Feasibility study (NCT04402333) completed recently at the Royal Surrey County Hospital in Guildford showed significantly enhanced recovery with short length of stay and reduced blood loss enabling faster recommencement of chemotherapy in women with advanced disease undergoing robotic surgery compared to open surgery (requiring a cut in the abdomen).

In the current proposed study funded by Intuitive Foundation and GRACE Charity, the investigators will establish the feasibility of conducting a randomised controlled trial and collect data from three hospital sites to inform a future phase 3 randomised controlled trial. The aim will be to to improve patient experience, access to surgery, recovery, reduce morbidity and reduce time to chemotherapy by incorporating robotic cytoreductive surgery into the ovarian cancer treatment pathway for women with a pelvic mass </=8cm

DETAILED DESCRIPTION:
Hypothesis: in selected cases of epithelial ovarian cancer (EOC), following neoadjuvant chemotherapy, robotic surgery is safe and acceptable, facilitates maximal debulking surgery and is associated with improved patient outcomes.

MIRRORS- RCT Pilot is a Randomised controlled trial (RCT) to establish whether; the MIRRORS protocol can operate successfully as an RCT at other sites, that patients are willing to be recruited and randomised, before commencing a national multicentre trial. The aim is to provide proof of the concept that a larger adequately powered multi-centre RCT is feasible.

All Women with Stage 3c or greater EOC with a pelvic mass ≤8cm will be identified at diagnosis from the first MDT discussion. All patients will have a CT at presentation which will be used to screen women as suitable or not for inclusion. Potential eligible participants will be offered inclusion and provided with a participant information leaflet and study consent form to consider for at least 24 hours prior to review in clinic. Participants opting to participate will then undergo the consent process. They will sign the study consent form following discussion and have the opportunity to ask any questions they wish. This consent process will be carried out with an experienced member of the clinical team who is authorised, trained and competent to do so. Participants will then be asked to complete baseline questionnaires.

All screened patients will have the following anonymised basic information collected: date of birth, age, ethnicity, reason not eligible and reason for declining if eligible but declined.

Participants found to have progressive disease will not be offered cytoreductive surgery and will then be excluded from the trial.

Following recruitment to the study, eligible patients will be randomised by the PI or delegated member of the clinical investigating team at local sites in a 2:1 ratio MIRRORS vs standard management (SM) using the Sealed Envelope randomisation service. Eligibility and consent will be verified before each patient is randomised.

The two arms of the study are:

MIRRORS Protocol (Diagnostic Laparoscopy proceed to either robotic or open Interval cytoreductive surgery with conversion to open at any point should this be required to remove all visible disease).

Standard Open Interval Cytoreductive Surgery (Surgery will proceed directly with standard open interval cytoreductive surgery through an extended midline incision).

A surgery date will be arranged enabling all randomised patients are booked onto an appropriate theatre list (robotic or open) with an appropriately experienced surgeon. This will ensure that robotic resources and theatre time is not wasted.

Patients, surgeons and treating physicians will not be blinded to the treatment. However, the statistician conducting the analysis will be blinded to the treatment allocation.

At the second MDT review, following a CT performed after 2 or 3 cycles of chemotherapy, some randomised patients may have to be excluded from the study at this point; for example, due to disease progression. It is expected that the attrition will be balanced between treatment arms, but it is possible that given the relatively small numbers included in the study, there may be some imbalance in the groups at the end of the recruitment period.

As is standard practice, the surgery will be discussed in detail and informed consent for the surgery will be undertaken during the participant's next clinic visit. Consent will be re-confirmed on the morning of surgery. All participants who join the study are free to change their mind and withdraw at any time during the study. The decision will not affect their care in any way. The anonymised data that is collected up to the point of withdrawing can still be used in the final analysis of the results unless the participant does not wish this to happen. In such cases, the investigators will destroy the data. Participant's GP will be informed that they are taking part in the study. Consent for informing the GP forms part of the study consent form.

At the time of surgery, the standard practice for advanced ovarian cancer would be to proceed with an extended vertical cut on the abdomen to remove as much tumour as possible. Participants who are randomised to MIRRORS protocol will start the surgery with an initial laparoscopic assessment (a camera inserted though the belly button). This visual assessment is used to determine whether it is feasible to proceed with surgery robotically or whether full cytoreductive surgery to zero macroscopic residual disease would be best carried out through an open surgical approach.

If an open surgical approach is considered the optimum treatment for the patient and they have consented for this, then this will be done. If there is disease that cannot be removed robotically after starting by this route but can be removed via an open incision, the surgery will be converted to an open procedure if it is safe to do so. If there are any complications, the investigators may also need to convert to open surgery. Participants randomised to standard cytoreductive surgery will receive standard cytoreductive surgery through a midline laparotomy. The aim of the surgery whether by robotic or open is to remove all visible disease safely.

The study will involve questionnaires relating to recovery and quality of life and pain (these are established validated questionnaires); two are from the European Organisation for Research and Treatment of Cancer: "EORTC QLQ C30" & "EORTC QLQ OV28."Another is the Hospital Anxiety and Depression Scale which is used to assess levels of anxiety and depression that a person is experiencing. The EQ5D-5L questionnaire will be used to gather health economic data. Lastly, the investigators will be using a simple 11-point pain scale (0-10) to assess participants' pain. These questionnaires will be completed at certain time points starting at baseline and then following on from surgery.

Study participants will be followed up during their normal scheduled appointment times as per the standard of care. There will be no additional screening bloods or investigations beyond that already done as part of the surgical work up. If necessary, questionnaires can be completed by telephone (included in the study consent form).

Collection of PROMs will be carried out via the web-based portal using computers, tablet or smartphone devices. Data security is paramount with regular penetration testing. Information is stored according to national standards and no identifiable data is stored on internet connected devices/database. Account details are stored on internally hosted servers and authenticated through SSL encrypted web services. Upon consent, participants will be provided with a login to facilitate their access to the platform and offered access to the Database. This is provided in an email triggered by initial participant registration following initial contact in clinic.

The email provides a unique identifier which allows participants to access their assigned PROMs surveys for completion. Once the appropriate PROMs questionnaire is completed, the data is then stored in the platform; additionally, a notification is sent to the research team system so that they can confirm completion status for their participants. It is also possible for participants, who do not have an email address, to be recruited into the study by allocating them with a username and password, and if they don't have their own computer, they can use it with either a Trust computer, or a public device, e.g. in a library.

At least one face to face or remote proctoring session will be carried out to vet all new sites enrolled in MIRRORS RCT (pilot) to ensure that surgeons participating in the MIRRORS protocol arm of MIRRORS-RCT (pilot) are suitably experienced regarding the MIRRORS-Protocol and trained to do so.

The investigators aim to recruit 20 women across 3 sites within a 6-8 months recruitment window. The sample size is set pragmatically to give precision in the estimate of pre-defined feasibility criteria parameters such as consent rate, robotic operation rate and success rate (target debulking of R=0 achieved) with timely recruitment. Inclusion of 20 women is sufficient to ensure these rates can be estimated within a standard error of less than 10%, providing maximal confidence intervals for percentage estimates of +/-20%.

ELIGIBILITY:
Inclusion Criteria:

* Women with Stage IIIc-IVb epithelial ovarian cancer (EOC) (including cancer of the fallopian tube & peritoneum) undergoing neo-adjuvant chemotherapy
* Pelvic mass ≤8 cm on CT
* Age ≥18years

Exclusion Criteria:

* A Pelvic Mass >8cm
* Not Suitable for interval cytoreductive surgery.
* Lacks capacity to understand or complete trial documentation.
* Patients not suitable for laparoscopy,
* Specialist surgical support is required and open surgery is recommended by the speciality team involved.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment | Assessed at close of recruitment 6-8 months (recruitment period)
  Number of patients consented compared to the number offered inclusion expressed as a percentage.

SECONDARY OUTCOMES:
Rate of conversion to open surgery | through study completion, an average of 1 year
  Percentage of patients converted to open surgery after being deemed suitable for Robotic interval debulking surgery following initial diagnostic laparoscopy. Success criteria: Conversion to open surgery rate is less than 50% of the patient group deemed suitable for Robotic interval debulking surgery following initial diagnostic laparoscopy.
Blood loss | through study completion, an average of 1 year
  blood loss during surgery in mililitres
Maximal macroscopic cytoreduction rate (R=0 rate) | through study completion, an average of 1 year
  Percentage of patients undergoing MIRRORS protocol who achieve maximal macroscopic debulking i.e. no macroscopic residual disease present (R=0 rate) vs standard open interval cytoreductive surgery
Surgical complications | through study completion, an average of 1 year
  Intraoperative complications will be recorded. Post operative complications will be recorded and classified by Clavien-Dindo Classification. Success criteria: Complication rate is not higher for MIRRORS protocol compared to standard open interval cytoreductive surgery.
Length of stay | through study completion, an average of 1 year
  Days from operation date. Operation date=day 0
Days to chemotherapy | through study completion, an average of 1 year
  Days from operation date. Operation date=day 0
Cost of MIRRORS protocol vs standard interval cytoreductive surgery | through study completion, an average of 1 year
  Cost comparison focusing on resources used in hospital (surgery, length of stay, readmissions, outpatients, A&E) and in the community post discharge (primary and community care). Contacts with services and professionals will be converted to costs using validated national tariffs and NHS Reference costs.
  The primary health-related outcome for the economic analysis will be EQ-5D-5L, completed by participants at baseline and at each assessment point. Responses will be used to estimate the patients' health related quality of life (utility level) at each time point. This will be done by scoring the EQ-5D 5L using a validated national tariff. The utility scores will be integrated over time to provide the Quality Adjusted Life Years (QALYs), accrued by each participant over the duration of the trial.
  A comparison of the difference in costs and difference in QALYs over the trial period will be conducted using appropriate statistical tests to assess significance.
Pain assessment | through study completion, an average of 1 year
  Numeric rating scale (NRS11) 0 (no pain) - 10 (worst pain) At baseline and post-operatively; day 1, 3, 7, 10, 14, 21, 6 weeks
Quality of life following surgery (generic) expressed as QALY gain using EQ5D-5L | through study completion, an average of 1 year
  At baseline and post-operatively; day 1, 3, 7, 10, 14,21,6 weeks
Quality of life following surgery (cancer specific) | through study completion, an average of 1 year
  Assessed using patient reported outcome measure (PROM) European Organisation for Research and Treatment of Cancer (EORTC) Validated quality of life questionnaire (QLQ) for ovarian cancer (QLQ-C30/QLQ-OV28). This validated questionnaire consists of the core module and its associated ovarian cancer specific module. Completed at baseline, day 3 post surgery, 3 weeks post-surgery and 6 weeks post surgery.
Mental wellbeing | through study completion, an average of 1 year
  Hospital anxiety and depression scale (HADS) A (Anxiety) and D (Depression) scores are calculated separately. 0-7 = Normal, 8-10 = Borderline, 11-21 = Abnormal (case) Completed at baseline, day 3 post surgery, 3 weeks post-surgery and 6 weeks post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Butler-Manuel, MD, Principal Investigator — Royal Surrey NHS Foundation Trust
Locations (1):
- Royal Surrey NHS Foundation Trust, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated from this current study will be available upon request from Miss Christina Uwins (Christina.Uwins@nhs.net) as raw anonymised data for up to 5 years following completion and publication of the study. Participants have given their consent for the information collected from this study to be used to support other research in the future and to be shared anonymously with other researchers.
Time Frame: up to 5 years following completion and publication of the study
Access Criteria: The datasets generated from this current study will be available upon request from Miss Christina Uwins (Christina.Uwins@nhs.net) as raw anonymised data

REFERENCES:
- [Result] Uwins C, Assalaarachchi H, Bennett K, Read J, Tailor A, Crawshaw J, Chatterjee J, Ellis P, Skene SS, Michael A, Butler-Manuel S. MIRRORS: a prospective cohort study assessing the feasibility of robotic interval debulking surgery for advanced-stage ovarian cancer. Int J Gynecol Cancer. 2024 Jun 3;34(6):886-897. doi: 10.1136/ijgc-2024-005265. PMID 38561194